CLINICAL TRIAL: NCT06436963
Title: Narrative Medicine Combined With Case-Based Learning
Brief Title: Exploring the Application of Narrative Medicine Combined With Case-Based Learning in the Standardized Training of General Practice Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022KY815
Record Dates: First submitted 2024-05-17; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Narrative Medicine; Case-based Learning
MeSH Terms: conditions — Narrative Medicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- narrative medicine training combined with CBL training (Experimental): The experimental group received narrative medicine training combined with CBL training
  Interventions: Behavioral: narrative medicine training combined with CBL training
- CBL training (Active Comparator): The control group received normal CBL training
  Interventions: Behavioral: CBL training

INTERVENTIONS:
Behavioral: narrative medicine training combined with CBL training — The experimental group received narrative medicine training combined with CBL training.
  Arms: narrative medicine training combined with CBL training
Behavioral: CBL training — The control group received normal CBL training.
  Arms: CBL training

SUMMARY:
This was a prospective, longitudinal, single-center nonrandomized controlled study. A total of 36 first- and second-year general practice residents of Zhejiang University School of Medicine were voluntarily enrolled in the experimental group. The remaining 9 residents served as a control group. The experimental group received narrative medicine training combined with CBL training. The control group received normal CBL training. None of the participants had previously had any training in narrative medicine. Teaching evaluation scores were measured for all subjects at baseline and 1 year after the training.

ELIGIBILITY:
Inclusion Criteria:

* first- and second-year general practice residents of Zhejiang University School of Medicine

Exclusion Criteria:

* third-year general practice residents of Zhejiang University School of Medicine

Ages: 24 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction Survey of Residents in the Experimental Group | 12 months
  The satisfaction survey was divided into five levels, ranging from "strongly agree" to "strongly disagree". The higher percent of agree means better result.
Comparison of the SEGUE scale scores Between the Experimental Group and the Control Group | 12 months
  The SEGUE scale scores were generated by assigning a value of "1" for "yes", "0" for "no" and "0.5" for "cannot answer". High scores indicate stronger clinical communication skills.
Comparison of the JSE-S scale scores Between the Experimental Group and the Control Group | 12 months
  The JSE-S scale scores adopts a 7-point Likert scale ranging from "strongly disagree" to "strongly agree". The higher total score indicating a greater level of empathy.
Comparison of the SEGUE scale in Different Grades Before and After Training in the Experimental Group | 12 months
  The SEGUE scale scores were generated by assigning a value of "1" for "yes", "0" for "no" and "0.5" for "cannot answer". High scores indicate stronger clinical communication skills.
Comparison of the JSE-S scale in Different Grades Before and After Training in the Experimental Group | 12 months
  The JSE-S scale scores adopts a 7-point Likert scale ranging from "strongly disagree" to "strongly agree". The higher total score indicating a greater level of empathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No